CLINICAL TRIAL: NCT06164756
Title: Long-Term Follow-Up for Subjects Enrolled in the Ketamine for the Treatment of Depression in Parkinson's Disease (KET-PD) Trial
Brief Title: Long Term Follow Up KET-PD
Status: Enrolling by invitation | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Fox (Michael J.) Foundation for Parkinson's Research (Unknown); Yale School of Medicine Center for Brain Mind Health (Unknown)
Responsible Party: Principal Investigator, Sophie Holmes, Assistant Professor of Psychiatry, Yale University
Other Study IDs: 2000036071
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Parkinson's Disease; Depression
Keywords: Long Term Effect Ketamine Treatment
MeSH Terms: conditions — Parkinson Disease; Depression | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Experimental: Ketamine Infusion: Participants who received 6 infusions of ketamine (0.5 mg/kg IV, up to 60 mg total), administered over 40 minutes while on continuous cardiac monitoring and oximetry in the ongoing clinical trial (KET-PD trial; NCT04944017, HIC 2000030394)
  Interventions: Other: Cognitive Behavior Therapy (CBT); Other: Treatment As Usual (TAU)
- Placebo Comparator: Saline Infusion: Participants who received 6 infusions of placebo (saline IV), administered over 40 minutes while on continuous cardiac monitoring and oximetry in the ongoing clinical trial (KET-PD trial; NCT04944017, HIC 2000030394)
  Interventions: Other: Cognitive Behavior Therapy (CBT); Other: Treatment As Usual (TAU)

INTERVENTIONS:
Other: Cognitive Behavior Therapy (CBT) — Participants will receive 10 weeks of CBT
Other: Treatment As Usual (TAU) — Participants will receive standard of care treatment

SUMMARY:
The purpose of this study is to examine a) the longer-term effects of ketamine for treating depression in Parkinson's disease (PD) and b) the effects of CBT on maintaining the effects of ketamine.

DETAILED DESCRIPTION:
This is a roll-out study from the ongoing clinical trial (KET-PD trial; NCT04944017, HIC 2000030394). We will adopt an implementation science approach to have participants across ketamine and placebo groups in one of two arms: a) follow-up with treatment as usual (TAU) (at 3 and 6 months post-infusions); b) follow-up with 3 months of Cognitive Behavior Therapy (CBT) post-infusions, delivered remotely once per week, with follow-up assessments at 3 and 6 month timepoints. CBT is expected to have a superior sustained antidepressant response to the TAU follow-up group in both ketamine and placebo arms. We hypothesize that ketamine + CBT will show the most superior antidepressant response at follow-up.

ELIGIBILITY:
Eligibility is determined in the ongoing parent clinical trial (KET-PD trial; NCT04944017, HIC 2000030394).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of n=56 participants with PD and comorbid depression, age 40-80, are being recruited under the parent clinical trial. As of July 2023, 20 participants have been enrolled. We aim to follow-up our remaining participants longitudinally and, within this, to have 20 prospective participants receive CBT, such that we will have 20 participants in each follow-up arm (CBT vs. TAU), and ultimately 10 in each group (ketamine + CBT, ketamine + TAU, placebo + CBT, placebo + TAU).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-12-21 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Long-Term Change in Depression Severity | 3 Months and 6 Months
  Change in MADRS score following course of ketamine vs. placebo treatment at 3 and 6 month timepoints; and change in MADRS across treatment (ketamine/placebo) and follow-up (CBT/TAU) arms at 3 and 6 month timepoints. The scale used to measure depression severity is called The Montgomery-Åsberg Depression Rating Scale (MADRS). The MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. The overall score ranges from 0 to 60, higher MADRS score indicates more severe depression.

SECONDARY OUTCOMES:
Change in Apathy | 3 Months and 6 Months
  Changes in apathy determined by the Starkstein Apathy Scale (SAS) scale
Change in Anxiety | 3 Months and 6 Months
  Changes in anxiety determined by the State-Trait Anxiety Inventory (STAI) scale
Change in Parkinson's Symptom Severity | 3 Months and 6 Months
  Changes in Parkinson's symptom severity determined by the Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) scale
Change in Dyskinesia | 3 Months and 6 Months
  Changes in dyskinesia determined by the Unified Dyskinesia Rating Scale (UDysRS) scale
Change in Pain | 3 Months and 6 Months
  Changes in pain determined by the King's PD Pain Scale
Change in Fatigue | 3 Months and 6 Months
  Changes in fatigue determined by the Parkinson's Fatigue Scale (PFS)
Change in Anhedonia | 3 Months and 6 Months
  Changes in anhedonia determined by the Snaith-Hamilton Pleasure Scale (SHAPS)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie E. Holmes, PhD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No